CLINICAL TRIAL: NCT04930003
Title: Randomized, Blind, Placebo-controlled Phase- I Study and Randomized, Open Phase Phase-II Study of QazCoVac-P - COVID-19 Subunit Vaccine in Healthy Adult Volunteers From 18 Years Old and Elder
Brief Title: Reactogenicity, Safety and Immunogenicity of QazCoVac-P COVID-19 Vaccine
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Research Institute for Biological Safety Problems (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: QAZCOVAC-P-I/II-01/2020
Record Dates: First submitted 2021-02-22; First posted 2021-06-18 (Actual); Last update posted 2023-12-07 (Actual); Status verified 2023-12

CONDITIONS: Covid19; SARS-CoV Infection; Vaccine Adverse Reaction
Keywords: vaccine,; I/II phase,; safety,; immunogenicity,; QazCoVac-P
MeSH Terms: conditions — COVID-19; Severe Acute Respiratory Syndrome

STUDY DESIGN:
Intervention Model Description: Assignment
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Experimental: Phase 1 Adult-vaccine (A Sample, blind study) (Experimental): Group 1 (phase 1): 22 volunteers aged 18-50 years who will be the QazCoVac-P - COVID-19 twice spaced 21 days apart, intramuscularly, at a dose of 0.5 ml
  Interventions: Biological: QazCoVac-P -COVID-19 Subunit Vaccine
- Phase 1 Adult-Placebo (A Sample, blind study) (Placebo Comparator): Group 2 (phase 1): 22 volunteers aged 18-50 years who will be the Placebo twice spaced 21 days apart, intramuscularly, at a dose of 0.5 ml
  Interventions: Other: Placebo
- Phase 2 Adult-Vaccine, twice vaccination (An Open study) (Experimental): Group 3 (phase 2): 50 volunteers aged 18-50 years who will be the QazCoVac-P - COVID-19 twice spaced 21 days apart, intramuscularly, at a dose of 0.5 ml
  Interventions: Biological: QazCoVac-P -COVID-19 Subunit Vaccine
- Phase 2 Elderly-Vaccine, twice vaccination (An Open study) (Experimental): Group 4 (phase 2): 50 volunteers from 50 years old and elder who will be the QazCoVac-P - COVID-19 twice spaced 21 days apart, intramuscularly, at a dose of 0.5 ml
  Interventions: Biological: QazCoVac-P -COVID-19 Subunit Vaccine
- Phase 2 Adult-Vaccine, single vaccination (An Open study) (Experimental): Group 5 (phase 2): 50 volunteers aged 18-50 years who will be the QazCoVac-P - COVID-19 single vaccination, intramuscularly, at a dose of 0.5 ml
  Interventions: Biological: QazCoVac-P -COVID-19 Subunit Vaccine
- Phase 2 Elderly-Vaccine, single vaccination (An Open study) (Experimental): Group 6 (phase 2): 50 volunteers from 50 years old and elder who will be the QazCoVac-P - COVID-19 single vaccination, intramuscularly, at a dose of 0.5 ml
  Interventions: Biological: QazCoVac-P -COVID-19 Subunit Vaccine

INTERVENTIONS:
Biological: QazCoVac-P -COVID-19 Subunit Vaccine — QazCoVac-P (Subunit) Vaccine manufactured by Research Institute for Biological Safety Problems Republic of Kazakhstan
  Arms: Experimental: Phase 1 Adult-vaccine (A Sample, blind study); Phase 2 Adult-Vaccine, single vaccination (An Open study); Phase 2 Adult-Vaccine, twice vaccination (An Open study); Phase 2 Elderly-Vaccine, single vaccination (An Open study); Phase 2 Elderly-Vaccine, twice vaccination (An Open study)
Other: Placebo — The use of placebo: intramuscularly, twice, spaced 21 days apart, at a dose of 0.5 ml (22 volunteers)
  Arms: Phase 1 Adult-Placebo (A Sample, blind study)

SUMMARY:
Randomized, Blind, Placebo-controlled Phase- I Study and Randomized, Open Phase Phase-II Study of QazCoVac-P - COVID-19 Subunit Vaccine in Healthy Adult Volunteers From 18 Years Old and Elder

DETAILED DESCRIPTION:
Purpose of the Phase-I clinical study Evaluation of the safety, acceptability and immunogenicity of QazCoVac-P - COVID-19 Subunit vaccine when administered twice in healthy volunteers aged 18-50 years.

Purpose of the Phase-II clinical study Evaluation of the safety and immunogenicity of QazCoVac-P - COVID-19 Subunit vaccine with single and dual use in healthy volunteers aged 18 and above

ELIGIBILITY:
Inclusion Criteria:

* Availability of signed and dated informed consent of the volunteer to
* participate in the study
* Healthy male and female volunteers aged 18-50 and 50 and above.
* Ability and voluntary desire to independently keep records in the SelfObservation Diary, as well as to carry out all the repeated visits provided for in the study for control medical observation.
* The voluntary desire of females to use methods of reliable contraception throughout the entire period of their participation in the study.
* Negative results for IgM and IgG antibodies to SARS-CoV-2.
* Absence of COVID-19 diagnosis in history.
* Absence in the last 14 days of close contact with persons suspected of being infected with SARS-CoV-2, or persons whose diagnosis of COVID-19 has been confirmed with laboratory.
* Negative test results for human immunodeficiency virus (HIV), hepatitis B and hepatitis C.
* Negative PCR results for coronavirus SARS-CoV-2
* According to the results of a chest x-ray, there is no pathological process in the lungs.

Exclusion Criteria:

* Aggravated allergic history, drug intolerance, including hypersensitivity to any of the components of the study drug, as well as a history of serious adverse events during vaccine administration (such as allergic reactions, respiratory failure, angioedema, abdominal pain).
* Acute illness with a fever (body temperature ≥37.1°C) at the time of screening/randomization.
* Chronic alcohol and/or drug use in history.
* Clinically significant deviations from normal values during laboratory and/or imaging at screening.
* Women with a positive urine pregnancy test.
* Simultaneous treatment with immunosuppressive drugs, including corticosteroids (2 weeks) 4 weeks prior to study drug administration.
* Acute or chronic clinically significant lesions of the lungs, cardiovascular system, gastrointestinal tract, liver, blood system, skin, endocrine, neurological and psychiatric diseases or impaired renal function (asthma, diabetes, thyroid disease, arrhythmia, myocardial infarction, severe hypertension not controlled by drugs, etc.), identified based on medical history, physical examination or clinical laboratory tests that, according to the researcher, may affect the study result.
* Disruption of platelets or other blood clotting disorders, which may cause contraindications to intramuscular administration.
* Leukemia or neoplasm in history.
* Persons with autoimmune diseases.
* Volunteers who received antiviral drugs, immunoglobulin's or blood transfusions or any other investigational drug within 4 weeks prior to study drug administration;
* Volunteers who received anti-inflammatory drugs 2 days before study drug
* administration;
* Participation in any other clinical research within the last 3 months;
* Volunteers with a concern that they will not comply with the study requirements, or persons with severe physical or mental disabilities that may affect the completion of the study;
* Negative PCR results for coronavirus SARS-CoV-2;
* According to the results of a chest x-ray, there is no pathological process in the lungs;
* Voluntary refusal to study;
* Vulnerable Volunteers of research.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 244 (Actual)
Dates: Start 2021-06-15 (Actual); Primary Completion 2021-12-15 (Actual); Study Completion 2021-12-15 (Actual)

PRIMARY OUTCOMES:
Frequency of adverse events up to seven days after immunization | Seven days after each immunization
  Frequency of adverse reaction in the seven days following each immunization per age group
Frequency of adverse events up to 21 days after immunization | 21 days after each immunization
  Frequency of adverse reaction in the 21 days following each immunization per age group
The proportion of volunteers with increased levels of the immune response of specific neutralizing antibody titers in ELISA following the vaccination, compared with a placebo | at days 0, 21, 27, 42, 90, 180
  The proportion of volunteers with changed levels of the immune response of specific neutralizing antibody titers in ELISA greater than ≥ 4 times compared with a placebo.

SECONDARY OUTCOMES:
Incidence of serious adverse events during the study | throughout the study, an average of 42 days
  Incidence of serious adverse events during the study.

OTHER OUTCOMES:
Cell-mediated immune profile | at days 0, 7, 21, 42
  Cellular immunity will be assessed by reliable (more than 2 standard deviations from the mean pre-vaccination level) increases in post-vaccination level (%) of CD4 + and CD8 + T-cells.

CONTACTS AND LOCATIONS:
Overall Officials: Kunsulu Zakarya, Ph.D., Study Chair — Research Institute for Biological Safety Problems
Locations (1):
- Research Institute for Biological Safety Problems Committee of Science of the Ministry of Education and Science of the Republic of Kazakhstan, Gvardeyskiy, Jambul, Kazakhstan